CLINICAL TRIAL: NCT04438434
Title: Evaluation of a Filming Formulation of Hydrogen Peroxide and Hyaluronic Acid (BMG0703) in Promoting the Healing of Post-extraction Sites, Compared to Placebo and 0.2% Chlorhexidine. A Randomised Controlled Clinical Trial.
Brief Title: Evaluation of Hydrogen Peroxide and Hyaluronic Acid (BMG0703) in the Healing of Post-extraction Sites
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Collaborators: BMG Pharma (Industry)
Responsible Party: Principal Investigator, Chiara Occhipinti, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orto_BMG0703_WIS_June_2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Impacted Third Molar Tooth; Healing Surgical Wounds
Keywords: Impacted Third Molar Tooth; Surgical wound healing; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The products will be packaged in such a way that they are not recognizable either by the operator or by the patient. Each package will be assigned a number that in turn will refer to the type of the product. The association between the number and type of the product will be collected by another operator on the basis of the association carried out by a dedicated software. The operator who will deliver the product will be informed about the type only at the end of the treatment.
  The data will be collected in pseudonymised form and inserted into a dedicated database in order to carry out the statistical analysis provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrogen Peroxide and Hyaluronic acid mouthwash (BMG0703) (Experimental): The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  The treatment to be evaluated involves mouth rinsing with 10 ml of BMG0703 three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to the product will be advised to discontinue its use, and seek medical advice.
  Interventions: Drug: Filming Formulation of Hydrogen Peroxide and Hyaluronic Acid
- Chlorhexidine 0.2% mouthwash (Active Comparator): The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  Subjects in this group are to use Chlorhexidine 0.2% mouthwash as an active comparator; 10 ml three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to Chlorhexidine will be advised to discontinue its use, and seek medical advice.
  Interventions: Drug: Chlorhexidine mouthwash
- Placebo product (Placebo Comparator): The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  Subjects in this group are to use a placebo product, and will be instructed to use 10 ml for mouth rinsing three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to the product will be advised to discontinue its use, and seek medical advice.
  Interventions: Other: Placebo product

INTERVENTIONS:
Drug: Filming Formulation of Hydrogen Peroxide and Hyaluronic Acid — The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  The treatment to be evaluated involves mouth rinsing with 10 ml of BMG0703 three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to the product will be advised to discontinue its use, and seek medical advice.
  Other Names: BMG0703
  Arms: Hydrogen Peroxide and Hyaluronic acid mouthwash (BMG0703)
Drug: Chlorhexidine mouthwash — The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  Subjects in this group are to use Chlorhexidine 0.2% mouthwash as an active comparator; 10 ml three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to Chlorhexidine will be advised to discontinue its use, and seek medical advice.
  Other Names: Chlorhexidine 0.2%
  Arms: Chlorhexidine 0.2% mouthwash
Other: Placebo product — The enrolled subjects will be examined and treated by specialized medical personnel.
  The extraction will be carried out by an experienced operator and will follow the standard guidelines for the extraction of impacted teeth. Once the tooth has been removed, a suture with detached stitches using silk thread 3/0 will be applied.
  From a pharmacological point of view, the patient will be prescribed antibiotic therapy (Amoxicillin 1g) to be administered twice daily for seven days, analgesic/anti-inflammatory therapy with NSAIDs (e.g. Synflex 550 mg/Brufen 800 mg) are to be used for a maximum of twice daily.
  Subjects in this group are to use a placebo product, and will be instructed to use 10 ml for mouth rinsing three times daily, after meals and after normal oral hygiene procedures, for one week (date of the follow-up visit).
  Patients with allergic reactions or hypersensitivity to the product will be advised to discontinue its use, and seek medical advice.
  Other Names: Placebo
  Arms: Placebo product

SUMMARY:
A clinical study to evaluate the efficacy and safety of a mouthwash containing Hydrogen Peroxide, Sodium Hyaluronate and Glycine in the healing of post-extraction sites of wisdom teeth by film forming action.

DETAILED DESCRIPTION:
57 subjects, with an indication for a third molar extraction, will be enrolled in the study. Participants selection will take place at the IRCCS "Ca" Granda Ospedale Maggiore Policlinico of Milan - UOC Surgery Maxillo Facial and Dentistry where the internship activity of the Degree Course in Dentistry and Dental Prosthetics, Dental Hygiene and the School of Specialization in Orthodontics of the University of Milan is held.

Subsequently, subjects will be equally divided and randomly assigned into the test or control groups. Assessment of outcomes will be carried out at a distance of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of informed consent
* Need to carry out extraction of a third molar in total or partial impaction

Exclusion Criteria:

* subjects suffering from HIV
* subjects suffering from hepatitis
* serious systemic diseases preventing the use of specific dental therapies
* acute and/or chronic infectious diseases
* inability to provide consent

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Healing Index (Laundry-Turnbull and Howley, modified by Pippi and coll. in 2015) | 7 days
  For evaluation of healing, the Laundry-Turnbull and Howley index will be used, considering the changes made by Pippi and coll. in 2015. In particular, seven parameters will be evaluated; a value of 1 or 0 will be assigned to each of these parameters; the sum of the values will indicate the degree of healing to be subsequently compared between the different groups.
  In particular, seven parameters will be assessed, to each of which a value of 1 or 0 will be assigned. The sum of the values will indicate the degree of healing to be compared between the different groups.
  These seven parameters are: redness of mucosa, granulation tissue, suppuration, swelling, re-epithelialization, bleeding, pain on palpation.
  Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giampietro Farronato, Professor, Principal Investigator — University of Milan; Gianguido Cossellu, Fellow, Principal Investigator — University of Milan
Locations (1):
- UOC Maxillofacial Surgery and Odontology, University of Milan, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data available upon request

REFERENCES:
- [Background] Rahban SR, Garner WL. Fibroproliferative scars. Clin Plast Surg. 2003 Jan;30(1):77-89. doi: 10.1016/s0094-1298(02)00069-x. PMID 12636218
- [Background] Araujo MG, Silva CO, Misawa M, Sukekava F. Alveolar socket healing: what can we learn? Periodontol 2000. 2015 Jun;68(1):122-34. doi: 10.1111/prd.12082. PMID 25867983
- [Background] Cosyn J, Sabzevar MM. Subgingival chlorhexidine varnish administration as an adjunct to same-day full-mouth root planing. II. Microbiological observations. J Periodontol. 2007 Mar;78(3):438-45. doi: 10.1902/jop.2007.060222. PMID 17335366
- [Background] Lee CT, Zhang S, Leung YY, Li SK, Tsang CC, Chu CH. Patients' satisfaction and prevalence of complications on surgical extraction of third molar. Patient Prefer Adherence. 2015 Feb 10;9:257-63. doi: 10.2147/PPA.S76236. eCollection 2015. PMID 25709411
- [Background] Bouloux GF, Steed MB, Perciaccante VJ. Complications of third molar surgery. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):117-28, vii. doi: 10.1016/j.coms.2006.11.013. PMID 18088870
- [Derived] Boccalari E, Khijmatgar S, Occhipinti C, Del Fabbro M, Inchingolo F, Tartaglia GM. Effect of hydrogen peroxide and hyaluronic acid in mouth rinse after third molar extraction: a triple-blind parallel randomized controlled clinical trial. Eur Rev Med Pharmacol Sci. 2024 Jul;28(13):3946-3957. doi: 10.26355/eurrev_202407_36527. PMID 39012233